CLINICAL TRIAL: NCT04930445
Title: An Open Label, Observational, Prospective Registry of Participants With Sickle Cell Disease (SCD) Treated With Oxbryta® (Voxelotor)
Brief Title: Oxbryta® Product Registry An Observational Study Designed to Evaluate the Effect of Oxbryta in Individuals With SCD
Acronym: PROSPECT
Status: Terminated | Type: Observational
Why Stopped: Emerging clinical data evaluated by Pfizer and shared with regulatory authorities indicates that the risk profile of voxelotor in people with SCD exceeds the benefits observed in previously generated global research, and requires further assessment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: GBT440-4R2; C5341019 (Other: Alias Study Number)
Record Dates: First submitted 2021-06-04; First posted 2021-06-18 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Registry Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Oxbryta Product Registry
  Interventions: Drug: Oxbryta® (voxelotor) 500mg Tablets

INTERVENTIONS:
Drug: Oxbryta® (voxelotor) 500mg Tablets — Participants will receive treatment with Oxbryta as prescribed by their physician, as part of their usual care. Participants will be treated and evaluated per standard of care (SOC) and at the physician's discretion. There are no pre-defined treatment requirements.
  Other Names: Voxelotor; Oxbryta®

SUMMARY:
This registry is an observational study designed to evaluate the effect of Oxbryta in individuals with SCD in a real-world setting.

DETAILED DESCRIPTION:
The study will be conducted at approximately 45 sites in the United States.

This registry is an observational study to evaluate the effects of Oxbryta in individuals with SCD. Any participant who is currently taking Oxbryta, or has been prescribed and will initiate treatment with Oxbryta, is eligible to participate. Eligible participants will receive treatment with Oxbryta as prescribed by their physician, as part of their usual care. Participants will be treated and evaluated per standard of care (SOC) and at the physician's discretion. This study will collect data that are recorded in the participants' medical records and other secondary data sources. Study data will be collected at regular intervals and entered in case report forms (CRFs) via an electronic data capture (EDC) system by the study staff. Participants will be considered to be on study for up to 5 years after their first dose of Oxbryta treatment, or until they withdraw their consent to participate, or are discontinued from the study. Treatment, including interruptions and restarting treatment, will continue at the discretion of the treating physician, and there are no pre-defined treatment requirements. Participants may receive any additional medications prescribed by their treating physician, or have any medical interventions that are deemed appropriate by the treating physician or study doctor. The participant or treating physician may discontinue Oxbryta at any time. Participants who discontinue treatment with Oxbryta earlier than 5 years will continue to be followed on study to collect clinical and quality of life (QoL) outcomes for up to 5 years after their first dose of Oxbryta treatment. Participant safety and tolerability will be assessed throughout the study data collection period by the study doctor and reported to the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet all the following criteria will be eligible for enrollment:

  1. Willing and able to provide written informed consent (aged ≥ 18 years), parental/ guardian consent and participant assent (aged ≥ 12 to <18 years) per local regulations, or pediatric participants (aged 4 to <12 years) with parental/guardian consent per Institutional Review Board (IRB) policy and requirements, consistent with ICH guidelines
  2. Male or female participants with documented diagnosis of sickle cell disease (all genotypes)
  3. Undergoing treatment with Oxbryta according to the Oxbryta USPI

Exclusion Criteria:

* Participants meeting any of the following criteria will not be eligible for study enrollment:

  1. Current participation in an investigation clinical trial or expanded access program, in which the participant may be receiving voxelotor treatment.
  2. Medical, psychological, or behavioral condition that, in the opinion of the study doctor, would confound or interfere with evaluation of safety and/or effectiveness of the study drug, prevent compliance with the study protocol; preclude informed consent; or render the participant unable/unlikely to comply with the study procedures

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients at each participating study site who have been treated with Oxbryta will be considered for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (42):
  - University of South Alabama, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - Center for Inherited Blood Disorders, Orange, California
  - Bass Center for Childhood Cancer and Blood Disorders (Stanford Lucile Packard Children's Hospital), Palo Alto, California
  - Department of Pediatrics, Hematology section, Palo Alto, California
  - Stanford Children's Hospital, Palo Alto, California
  - University of Connecticut Health, Farmington, Connecticut
  - Nemours Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Health, Wilmington, Wilmington, Delaware
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Augusta University - Clinical Trials Office (clinic), Augusta, Georgia
  - Augusta University, Augusta, Georgia
  - University of Illinois at Chicago (UIC) Clinical Research Center, Chicago, Illinois
  - University of Illinois at Chicago (UIC) Sickle Cell Center, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System(UI Health), Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - University of Maryland Medical Center, College Park, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - ECU Health Medical Center Laboratory, Greenville, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - UPMC Montefiore Hospital, Pittsburgh, Pennsylvania
  - UPMC Sickle Cell Center, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Medical University of South Carolina Shawn Jenkins Women's and Children's Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Blood and Cancer Center at Dell Children's Medical Center, Austin, Texas
  - Dell Children's Medical Center, Austin, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - INOVA Health, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-4R2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 24 sites in the United States. The study was terminated as emerging clinical data indicated that the risk profile of Oxbryta (voxelotor) in participants with sickle cell disease (SCD) exceeded the benefits observed in previously generated global research and required further assessment. Screen failure was defined as participants who did not start or restart Oxbryta within six months of informed consent.
Pre-assignment Details: A total of 265 participants with SCD (all genotypes) aged greater than or equal to (>=) 5 years were enrolled in this study. Data was collected from participants medical records and other secondary data sources such as insurance and pharmacy claims. Participants were followed for up to 5 years after their first dose of Oxbryta treatment (irrespective of how long participants were on Oxbryta when they were enrolled in the study), or until they withdrew consent or were discontinued from study.
Groups:
- All Participants: Participants with SCD who were treated with Oxbryta in study C5341018 (NCT04930328) or were prescribed Oxbryta by their physician as part of their usual care were included.
Period: Overall Study
Arm/Group | All Participants
Started | 265
Treated | 260
Completed | 0
Not Completed | 265
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 1
Not completed — Study Terminated by Sponsor | 245
Not completed — Screen Failure | 8
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who met the inclusion/exclusion criteria and signed the inform consent, including screen failures (participants who did not receive Oxbryta within 6 months of the inform consent date).
Arm/Group | All Participants
Number analyzed (Participants) | 265
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.0 (14.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 240
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 246
  White | 6
  More than one race | 0
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin From Pre-Oxbryta Treatment (Baseline) Through Month 60 Post-Oxbryta
Description: The pre-Oxbryta (baseline) value was the latest measurement on or prior to the first dose of Oxbryta. Post-Oxbryta value was the measurement for multiple assessments at the same specific visit, the average was used.
Time Frame: Pre-Oxbryta (baseline) 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months post-Oxbryta
Population: FAS included all participants who met the inclusion/exclusion criteria and signed the inform consent, including screen failures (participants who did not receive Oxbryta within 6 months of the inform consent date). Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for specified time-points.
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | All Participants
Number analyzed (Participants) | 220
Grams per deciliter (g/dL)
  3 months Post-Oxbryta: number analyzed (Participants) | 215
  3 months Post-Oxbryta | 0.5 (1.33)
  6 months Post-Oxbryta: number analyzed (Participants) | 219
  6 months Post-Oxbryta | 0.6 (1.47)
  9 months Post-Oxbryta: number analyzed (Participants) | 205
  9 months Post-Oxbryta | 0.5 (1.45)
  12 months Post-Oxbryta: number analyzed (Participants) | 209
  12 months Post-Oxbryta | 0.6 (1.36)
  18 months Post-Oxbryta | 0.7 (1.35)
  24 months Post-Oxbryta: number analyzed (Participants) | 184
  24 months Post-Oxbryta | 0.6 (1.46)
  30 months Post-Oxbryta: number analyzed (Participants) | 155
  30 months Post-Oxbryta | 0.5 (1.62)
  36 months Post-Oxbryta: number analyzed (Participants) | 122
  36 months Post-Oxbryta | 0.6 (1.62)
  42 months Post-Oxbryta: number analyzed (Participants) | 103
  42 months Post-Oxbryta | 0.4 (1.48)
  48 months Post-Oxbryta: number analyzed (Participants) | 77
  48 months Post-Oxbryta | 0.7 (1.47)
  54 months Post-Oxbryta: number analyzed (Participants) | 41
  54 months Post-Oxbryta | 0.1 (1.68)
  60 months Post-Oxbryta: number analyzed (Participants) | 8
  60 months Post-Oxbryta | -0.2 (1.36)

2. Primary Outcome: Change in Percent Reticulocyte Count From Pre-Oxbryta Treatment (Baseline) Through Month 60 Post-Oxbryta
Description: as for outcome 1
Time Frame: Pre-Oxbryta (baseline) 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months post-Oxbryta
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | All Participants
Number analyzed (Participants) | 169
Percentage of reticulocytes
  3 months Post-Oxbryta: number analyzed (Participants) | 164
  3 months Post-Oxbryta | -0.9 (5.50)
  6 months Post-Oxbryta: number analyzed (Participants) | 158
  6 months Post-Oxbryta | -1.1 (6.01)
  9 months Post-Oxbryta: number analyzed (Participants) | 147
  9 months Post-Oxbryta | -1.1 (5.97)
  12 months Post-Oxbryta: number analyzed (Participants) | 163
  12 months Post-Oxbryta | -1.2 (6.34)
  18 months Post-Oxbryta | -1.6 (6.69)
  24 months Post-Oxbryta: number analyzed (Participants) | 143
  24 months Post-Oxbryta | -0.7 (6.32)
  30 months Post-Oxbryta: number analyzed (Participants) | 118
  30 months Post-Oxbryta | -1.0 (6.92)
  36 months Post-Oxbryta: number analyzed (Participants) | 86
  36 months Post-Oxbryta | -1.3 (7.04)
  42 months Post-Oxbryta: number analyzed (Participants) | 77
  42 months Post-Oxbryta | -0.2 (7.45)
  48 months Post-Oxbryta: number analyzed (Participants) | 52
  48 months Post-Oxbryta | 0.2 (6.70)
  54 months Post-Oxbryta: number analyzed (Participants) | 36
  54 months Post-Oxbryta | -0.3 (6.59)
  60 months Post-Oxbryta: number analyzed (Participants) | 7
  60 months Post-Oxbryta | 1.9 (3.84)

3. Primary Outcome: Change in Absolute Reticulocyte Count From Pre-Oxbryta Treatment (Baseline) Through Month 60 Post-Oxbryta
Description: as for outcome 1
Time Frame: Pre-Oxbryta (baseline) 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months post-Oxbryta
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | All Participants
Number analyzed (Participants) | 136
10^9 cells/Liter
  3 months Post-Oxbryta | 1.5 (134.05)
  6 months Post-Oxbryta: number analyzed (Participants) | 128
  6 months Post-Oxbryta | -4.1 (137.59)
  9 months Post-Oxbryta: number analyzed (Participants) | 123
  9 months Post-Oxbryta | -15.6 (188.54)
  12 months Post-Oxbryta: number analyzed (Participants) | 126
  12 months Post-Oxbryta | 2.4 (130.76)
  18 months Post-Oxbryta: number analyzed (Participants) | 128
  18 months Post-Oxbryta | -17.8 (175.27)
  24 months Post-Oxbryta: number analyzed (Participants) | 108
  24 months Post-Oxbryta | 31.4 (242.25)
  30 months Post-Oxbryta: number analyzed (Participants) | 93
  30 months Post-Oxbryta | 0.1 (134.67)
  36 months Post-Oxbryta: number analyzed (Participants) | 63
  36 months Post-Oxbryta | -15.3 (228.15)
  42 months Post-Oxbryta: number analyzed (Participants) | 55
  42 months Post-Oxbryta | 2.7 (142.52)
  48 months Post-Oxbryta: number analyzed (Participants) | 37
  48 months Post-Oxbryta | 4.4 (119.59)
  54 months Post-Oxbryta: number analyzed (Participants) | 23
  54 months Post-Oxbryta | 3.3 (140.03)
  60 months Post-Oxbryta: number analyzed (Participants) | 3
  60 months Post-Oxbryta | 21.7 (93.55)

4. Primary Outcome: Change in Bilirubin (Total, Direct and Indirect) Level From Pre-Oxbryta Treatment (Baseline) Through Month 60 Post-Oxbryta
Description: The pre-Oxbryta (baseline) value was the latest measurement on or prior to the first dose of Oxbryta. Post-Oxbryta value was the measurement for multiple assessments at the same specific visit, the average was used. Abbreviations used: overall number of participants analyzed=N and Number analyzed= n
Time Frame: Pre-Oxbryta (baseline) 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months post-Oxbryta
Population: FAS included all participants who met the inclusion/exclusion criteria and signed inform consent, including screen failures (participants who did not receive Oxbryta within 6 months of inform consent date). Here, 'N'=number of participants evaluable for this outcome measure and 'n'=participants evaluable for specified time-points. Indirect bilirubin data for month 54 and 60 was not collected as data collection was not mandatory for laboratory parameters since it is a non-interventional study.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | All Participants
Number analyzed (Participants) | 194
milligrams per deciliter (mg/dL)
  3 months Post-Oxbryta: Direct: number analyzed (Participants) | 74
  3 months Post-Oxbryta: Direct | 0.0 (0.57)
  6 months Post-Oxbryta: Direct: number analyzed (Participants) | 75
  6 months Post-Oxbryta: Direct | -0.1 (0.46)
  9 months Post-Oxbryta: Direct: number analyzed (Participants) | 65
  9 months Post-Oxbryta: Direct | 0.0 (0.35)
  12 months Post-Oxbryta: Direct: number analyzed (Participants) | 64
  12 months Post-Oxbryta: Direct | 0.1 (1.22)
  18 months Post-Oxbryta: Direct: number analyzed (Participants) | 82
  18 months Post-Oxbryta: Direct | 0.1 (1.57)
  24 months Post-Oxbryta: Direct: number analyzed (Participants) | 66
  24 months Post-Oxbryta: Direct | 0.1 (1.01)
  30 months Post-Oxbryta: Direct: number analyzed (Participants) | 54
  30 months Post-Oxbryta: Direct | 0.2 (0.81)
  36 months Post-Oxbryta: Direct: number analyzed (Participants) | 38
  36 months Post-Oxbryta: Direct | -0.1 (0.31)
  42 months Post-Oxbryta: Direct: number analyzed (Participants) | 35
  42 months Post-Oxbryta: Direct | 0.1 (0.62)
  48 months Post-Oxbryta: Direct: number analyzed (Participants) | 25
  48 months Post-Oxbryta: Direct | -0.1 (0.37)
  54 months Post-Oxbryta: Direct: number analyzed (Participants) | 15
  54 months Post-Oxbryta: Direct | -0.1 (0.28)
  60 months Post-Oxbryta: Direct: number analyzed (Participants) | 4
  60 months Post-Oxbryta: Direct | -0.1 (0.37)
  3 months Post-Oxbryta: Indirect: number analyzed (Participants) | 27
  3 months Post-Oxbryta: Indirect | -0.4 (1.19)
  6 months Post-Oxbryta: Indirect: number analyzed (Participants) | 27
  6 months Post-Oxbryta: Indirect | -0.3 (1.28)
  9 months Post-Oxbryta: Indirect: number analyzed (Participants) | 28
  9 months Post-Oxbryta: Indirect | 0.0 (2.23)
  12 months Post-Oxbryta: Indirect: number analyzed (Participants) | 23
  12 months Post-Oxbryta: Indirect | -0.5 (1.22)
  18 months Post-Oxbryta: Indirect: number analyzed (Participants) | 28
  18 months Post-Oxbryta: Indirect | 0.4 (2.64)
  24 months Post-Oxbryta: Indirect: number analyzed (Participants) | 23
  24 months Post-Oxbryta: Indirect | 0.2 (1.23)
  30 months Post-Oxbryta: Indirect: number analyzed (Participants) | 17
  30 months Post-Oxbryta: Indirect | 0.2 (1.40)
  36 months Post-Oxbryta: Indirect: number analyzed (Participants) | 11
  36 months Post-Oxbryta: Indirect | 0.0 (0.97)
  42 months Post-Oxbryta: Indirect: number analyzed (Participants) | 6
  42 months Post-Oxbryta: Indirect | -0.4 (0.78)
  48 months Post-Oxbryta: Indirect: number analyzed (Participants) | 5
  48 months Post-Oxbryta: Indirect | -0.1 (1.45)
  54 months Post-Oxbryta: Indirect: number analyzed (Participants) | 0
  60 months Post-Oxbryta: Indirect: number analyzed (Participants) | 0
  3 months Post-Oxbryta: Total: number analyzed (Participants) | 184
  3 months Post-Oxbryta: Total | -0.5 (1.71)
  6 months Post-Oxbryta: Total: number analyzed (Participants) | 189
  6 months Post-Oxbryta: Total | -0.5 (1.97)
  9 months Post-Oxbryta: Total: number analyzed (Participants) | 171
  9 months Post-Oxbryta: Total | -0.2 (2.76)
  12 months Post-Oxbryta: Total: number analyzed (Participants) | 177
  12 months Post-Oxbryta: Total | -0.4 (2.66)
  18 months Post-Oxbryta: Total | -0.5 (2.24)
  24 months Post-Oxbryta: Total: number analyzed (Participants) | 164
  24 months Post-Oxbryta: Total | -0.4 (2.27)
  30 months Post-Oxbryta: Total: number analyzed (Participants) | 138
  30 months Post-Oxbryta: Total | -0.3 (2.10)
  36 months Post-Oxbryta: Total: number analyzed (Participants) | 101
  36 months Post-Oxbryta: Total | -0.5 (2.48)
  42 months Post-Oxbryta: Total: number analyzed (Participants) | 92
  42 months Post-Oxbryta: Total | -0.5 (2.90)
  48 months Post-Oxbryta: Total: number analyzed (Participants) | 68
  48 months Post-Oxbryta: Total | -0.8 (2.59)
  54 months Post-Oxbryta: Total: number analyzed (Participants) | 36
  54 months Post-Oxbryta: Total | -0.6 (2.56)
  60 months Post-Oxbryta: Total: number analyzed (Participants) | 6
  60 months Post-Oxbryta: Total | -0.1 (1.33)

5. Primary Outcome: Change in Iron Overload (Ferritin Levels) From Pre-Oxbryta Treatment (Baseline) Through Month 60 Post-Oxbryta
Description: as for outcome 1
Time Frame: Pre-Oxbryta (baseline) 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months post-Oxbryta
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms per liter
Arm/Group | All Participants
Number analyzed (Participants) | 84
Micrograms per liter
  3 months Post-Oxbryta: number analyzed (Participants) | 69
  3 months Post-Oxbryta | 74.0 (1696.32)
  6 months Post-Oxbryta: number analyzed (Participants) | 71
  6 months Post-Oxbryta | 105.2 (1995.71)
  9 months Post-Oxbryta: number analyzed (Participants) | 69
  9 months Post-Oxbryta | -60.7 (2200.70)
  12 months Post-Oxbryta: number analyzed (Participants) | 62
  12 months Post-Oxbryta | 136.9 (1614.56)
  18 months Post-Oxbryta | 148.0 (1973.60)
  24 months Post-Oxbryta: number analyzed (Participants) | 75
  24 months Post-Oxbryta | 94.0 (2111.95)
  30 months Post-Oxbryta: number analyzed (Participants) | 58
  30 months Post-Oxbryta | -248.1 (1761.49)
  36 months Post-Oxbryta: number analyzed (Participants) | 45
  36 months Post-Oxbryta | -220.5 (1765.71)
  42 months Post-Oxbryta: number analyzed (Participants) | 41
  42 months Post-Oxbryta | 667.5 (2577.61)
  48 months Post-Oxbryta: number analyzed (Participants) | 31
  48 months Post-Oxbryta | 896.7 (3142.23)
  54 months Post-Oxbryta: number analyzed (Participants) | 21
  54 months Post-Oxbryta | 1672.8 (3975.50)
  60 months Post-Oxbryta: number analyzed (Participants) | 4
  60 months Post-Oxbryta | 4512.5 (5500.90)

6. Primary Outcome: Change in Iron Overload as Measured by T2-weighted Magnetic Resonance Imaging (MRI) From Pre-Oxbryta Treatment (Baseline) Through Month 60 Post-Oxbryta
Description: as for outcome 1
Time Frame: Pre-Oxbryta (baseline) up to 60 months post-Oxbryta
Population: No data was not collected for this outcome measure as the information regarding iron overload as measured by T2-weighted MRI was not available in the medical record for any of the participants.
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Primary Outcome: Change in Serum Creatinine Level From Pre-Oxbryta Treatment (Baseline) Through Month 60 Post-Oxbryta
Description: as for outcome 1
Time Frame: Pre-Oxbryta (baseline) 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months post-Oxbryta
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | All Participants
Number analyzed (Participants) | 206
milligrams per deciliter (mg/dL)
  3 months Post-Oxbryta: number analyzed (Participants) | 199
  3 months Post-Oxbryta | 0.0 (0.37)
  6 months Post-Oxbryta: number analyzed (Participants) | 195
  6 months Post-Oxbryta | 0.0 (0.46)
  9 months Post-Oxbryta: number analyzed (Participants) | 183
  9 months Post-Oxbryta | 0.1 (0.60)
  12 months Post-Oxbryta: number analyzed (Participants) | 187
  12 months Post-Oxbryta | 0.0 (0.37)
  18 months Post-Oxbryta | 0.1 (0.43)
  24 months Post-Oxbryta: number analyzed (Participants) | 176
  24 months Post-Oxbryta | 0.1 (0.51)
  30 months Post-Oxbryta: number analyzed (Participants) | 146
  30 months Post-Oxbryta | 0.2 (0.60)
  36 months Post-Oxbryta: number analyzed (Participants) | 115
  36 months Post-Oxbryta | 0.2 (0.92)
  42 months Post-Oxbryta: number analyzed (Participants) | 100
  42 months Post-Oxbryta | 0.3 (1.04)
  48 months Post-Oxbryta: number analyzed (Participants) | 70
  48 months Post-Oxbryta | 0.1 (0.52)
  54 months Post-Oxbryta: number analyzed (Participants) | 38
  54 months Post-Oxbryta | 0.4 (1.17)
  60 months Post-Oxbryta: number analyzed (Participants) | 8
  60 months Post-Oxbryta | 0.1 (0.25)

8. Primary Outcome: Change in Albumin Creatinine Ratio (ACR) From Pre-Oxbryta Treatment (Baseline) Through Month 54 Post-Oxbryta
Description: as for outcome 1
Time Frame: Pre-Oxbryta (baseline) 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 months post-Oxbryta
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram per gram
Arm/Group | All Participants
Number analyzed (Participants) | 20
Milligram per gram
  3 months Post-Oxbryta: number analyzed (Participants) | 17
  3 months Post-Oxbryta | 67.5 (451.66)
  6 months Post-Oxbryta: number analyzed (Participants) | 15
  6 months Post-Oxbryta | -42.1 (137.70)
  9 months Post-Oxbryta: number analyzed (Participants) | 13
  9 months Post-Oxbryta | 59.6 (129.88)
  12 months Post-Oxbryta: number analyzed (Participants) | 13
  12 months Post-Oxbryta | -32.1 (158.67)
  18 months Post-Oxbryta | 125.2 (330.70)
  24 months Post-Oxbryta: number analyzed (Participants) | 17
  24 months Post-Oxbryta | 7.7 (178.23)
  30 months Post-Oxbryta: number analyzed (Participants) | 14
  30 months Post-Oxbryta | 80.3 (164.48)
  36 months Post-Oxbryta: number analyzed (Participants) | 8
  36 months Post-Oxbryta | 14.4 (130.58)
  42 months Post-Oxbryta: number analyzed (Participants) | 11
  42 months Post-Oxbryta | 38.2 (96.87)
  48 months Post-Oxbryta: number analyzed (Participants) | 4
  48 months Post-Oxbryta | 273.3 (599.99)
  54 months Post-Oxbryta: number analyzed (Participants) | 3
  54 months Post-Oxbryta | 873.3 (1488.60)

9. Primary Outcome: Number of Participants According to Hemoglobinuria Results Post-Oxbryta
Description: Hemoglobinuria was defined as urine dipstick results positive for blood +1 or greater and <=2 red blood cells (RBC) by high power field. Number of participants according to hemoglobinuria results (none/negative, trace, 1+, 2+, 3+, other: large, moderate, small, small=0-3, hereditary persistence of fetal hemoglobin [HPF], missing) was reported in this outcome measure. Small corresponded to trace or 1+ on dipstick, medium indicated 2+, large indicated 3+ or higher on dipstick. The pre-Oxbryta (baseline) value was the latest measurement on or prior to the first dose of Oxbryta. Post-Oxbryta value was the measurement for multiple assessments at the same specific visit, the average was used.
Time Frame: Pre-Oxbryta (baseline) 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months post-Oxbryta
Population: FAS included all participants who met the inclusion/exclusion criteria and signed the inform consent, including screen failures (participants who did not receive Oxbryta within 6 months of the inform consent date).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 265
Participants
  Pre-Oxbryta: None/Negative | 22
  Pre-Oxbryta: Trace | 7
  Pre-Oxbryta: 1+ | 3
  Pre-Oxbryta: 2+ | 6
  Pre-Oxbryta: 3+ | 0
  Pre-Oxbryta: Other: Large | 3
  Pre-Oxbryta: Other: Moderate | 1
  Pre-Oxbryta: Other: Small | 0
  Pre-Oxbryta: Other: Small- 0-3 HPF | 0
  Pre-Oxbryta: Missing | 223
  3 months Post-Oxbryta: None/Negative | 7
  3 months Post-Oxbryta: Trace | 4
  3 months Post-Oxbryta: 1+ | 2
  3 months Post-Oxbryta: 2+ | 0
  3 months Post-Oxbryta: 3+ | 0
  3 months Post-Oxbryta: Other: Large | 0
  3 months Post-Oxbryta: Other: Moderate | 0
  3 months Post-Oxbryta: Other: Small | 1
  3 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  3 months Post-Oxbryta: Missing | 251
  6 months Post-Oxbryta: None/Negative | 12
  6 months Post-Oxbryta: Trace | 0
  6 months Post-Oxbryta: 1+ | 2
  6 months Post-Oxbryta: 2+ | 3
  6 months Post-Oxbryta: 3+ | 0
  6 months Post-Oxbryta: Other: Large | 0
  6 months Post-Oxbryta: Other: Moderate | 1
  6 months Post-Oxbryta: Other: Small | 0
  6 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  6 months Post-Oxbryta: Missing | 247
  9 months Post-Oxbryta: None/Negative | 8
  9 months Post-Oxbryta: Trace | 3
  9 months Post-Oxbryta: 1+ | 0
  9 months Post-Oxbryta: 2+ | 0
  9 months Post-Oxbryta: 3+ | 0
  9 months Post-Oxbryta: Other: Large | 0
  9 months Post-Oxbryta: Other: Moderate | 0
  9 months Post-Oxbryta: Other: Small | 0
  9 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  9 months Post-Oxbryta: Missing | 254
  12 months Post-Oxbryta: None/Negative | 11
  12 months Post-Oxbryta: Trace | 2
  12 months Post-Oxbryta: 1+ | 1
  12 months Post-Oxbryta: 2+ | 0
  12 months Post-Oxbryta: 3+ | 0
  12 months Post-Oxbryta: Other: Large | 0
  12 months Post-Oxbryta: Other: Moderate | 0
  12 months Post-Oxbryta: Other: Small | 1
  12 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  12 months Post-Oxbryta: Missing | 250
  18 months Post-Oxbryta: None/Negative | 18
  18 months Post-Oxbryta: Trace | 6
  18 months Post-Oxbryta: 1+ | 2
  18 months Post-Oxbryta: 2+ | 1
  18 months Post-Oxbryta: 3+ | 0
  18 months Post-Oxbryta: Other: Large | 0
  18 months Post-Oxbryta: Other: Moderate | 2
  18 months Post-Oxbryta: Other: Small | 0
  18 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  18 months Post-Oxbryta: Missing | 236
  24 months Post-Oxbryta: None/Negative | 17
  24 months Post-Oxbryta: Trace | 4
  24 months Post-Oxbryta: 1+ | 3
  24 months Post-Oxbryta: 2+ | 0
  24 months Post-Oxbryta: 3+ | 0
  24 months Post-Oxbryta: Other: Large | 0
  24 months Post-Oxbryta: Other: Moderate | 0
  24 months Post-Oxbryta: Other: Small | 2
  24 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  24 months Post-Oxbryta: Missing | 239
  30 months Post-Oxbryta: None/Negative | 16
  30 months Post-Oxbryta: Trace | 2
  30 months Post-Oxbryta: 1+ | 1
  30 months Post-Oxbryta: 2+ | 0
  30 months Post-Oxbryta: 3+ | 0
  30 months Post-Oxbryta: Other: Large | 0
  30 months Post-Oxbryta: Other: Moderate | 0
  30 months Post-Oxbryta: Other: Small | 0
  30 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  30 months Post-Oxbryta: Missing | 246
  36 months Post-Oxbryta: None/Negative | 13
  36 months Post-Oxbryta: Trace | 1
  36 months Post-Oxbryta: 1+ | 0
  36 months Post-Oxbryta: 2+ | 0
  36 months Post-Oxbryta: 3+ | 2
  36 months Post-Oxbryta: Other: Large | 2
  36 months Post-Oxbryta: Other: Moderate | 0
  36 months Post-Oxbryta: Other: Small | 0
  36 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  36 months Post-Oxbryta: Missing | 247
  42 months Post-Oxbryta: None/Negative | 12
  42 months Post-Oxbryta: Trace | 4
  42 months Post-Oxbryta: 1+ | 1
  42 months Post-Oxbryta: 2+ | 0
  42 months Post-Oxbryta: 3+ | 0
  42 months Post-Oxbryta: Other: Large | 1
  42 months Post-Oxbryta: Other: Moderate | 0
  42 months Post-Oxbryta: Other: Small | 1
  42 months Post-Oxbryta: Other: Small- 0-3 HPF | 1
  42 months Post-Oxbryta: Missing | 245
  48 months Post-Oxbryta: None/Negative | 12
  48 months Post-Oxbryta: Trace | 2
  48 months Post-Oxbryta: 1+ | 1
  48 months Post-Oxbryta: 2+ | 2
  48 months Post-Oxbryta: 3+ | 1
  48 months Post-Oxbryta: Other: Large | 0
  48 months Post-Oxbryta: Other: Moderate | 0
  48 months Post-Oxbryta: Other: Small | 0
  48 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  48 months Post-Oxbryta: Missing | 247
  54 months Post-Oxbryta: None/Negative | 8
  54 months Post-Oxbryta: Trace | 2
  54 months Post-Oxbryta: 1+ | 0
  54 months Post-Oxbryta: 2+ | 0
  54 months Post-Oxbryta: 3+ | 0
  54 months Post-Oxbryta: Other: Large | 1
  54 months Post-Oxbryta: Other: Moderate | 0
  54 months Post-Oxbryta: Other: Small | 1
  54 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  54 months Post-Oxbryta: Missing | 253
  60 months Post-Oxbryta: None/Negative | 1
  60 months Post-Oxbryta: Trace | 0
  60 months Post-Oxbryta: 1+ | 0
  60 months Post-Oxbryta: 2+ | 0
  60 months Post-Oxbryta: 3+ | 0
  60 months Post-Oxbryta: Other: Large | 0
  60 months Post-Oxbryta: Other: Moderate | 0
  60 months Post-Oxbryta: Other: Small | 0
  60 months Post-Oxbryta: Other: Small- 0-3 HPF | 0
  60 months Post-Oxbryta: Missing | 264

10. Primary Outcome: Change in Serum Cystatin C Results From Pre-Oxbryta Treatment (Baseline) Through Month 30 Post-Oxbryta
Description: as for outcome 1
Time Frame: Pre-Oxbryta (baseline) 3, 6, 12, 18, 24, 30 months post-Oxbryta
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | All Participants
Number analyzed (Participants) | 2
milligrams per liter (mg/L)
  3 months Post-Oxbryta: number analyzed (Participants) | 1
  3 months Post-Oxbryta | 0.1 (NA) — Standard deviation could not be estimated as a single participant was analyzed.
  6 months Post-Oxbryta | -0.1 (0.07)
  12 months Post-Oxbryta | 0.2 (0.07)
  18 months Post-Oxbryta | -0.2 (0.07)
  24 months Post-Oxbryta | 0.0 (0.11)
  30 months Post-Oxbryta | -0.1 (0.07)

11. Primary Outcome: Number of Participants According to Estimated Glomerular Filtration Rate (GFR) Results Post-Oxbryta
Description: Estimated GFR was calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. Number of participants according to estimated GFR results (stage 1 [G1] - GFR >=90 milliliter/minute [mL/min] per 1.73 square meters [m^2], stage 2 [G2] - GFR 60 to 89 mL/min per 1.73 m^2, stage 3a [G3a] - GFR 45 to 59 mL/min per 1.73 m^2, stage 3b [G3b] - GFR 30 to 44 mL/min per 1.73 m^2, stage 4 [G4] - GFR 15 to 29 mL/min per 1.73 m^2, stage 5 [G5] - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis, missing) was reported descriptively in this outcome measure. Stages 1 and 2 indicate mild damage, while stages 3 to 5 reflected progressive severity, leading to potential renal failure. The pre-Oxbryta (baseline) value was the latest measurement on or prior to the first dose of Oxbryta. Post-Oxbryta value was the measurement for multiple assessments at the same specific visit, the average was used.
Time Frame: Pre-Oxbryta (baseline) 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months post-Oxbryta
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 265
Participants
  Pre-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 63
  Pre-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 24
  Pre-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 8
  Pre-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 2
  Pre-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 3
  Pre-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 1
  Pre-Oxbryta: Missing | 164
  3 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 47
  3 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 21
  3 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 2
  3 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 1
  3 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 4
  3 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 1
  3 months Post-Oxbryta: Missing | 189
  6 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 51
  6 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 17
  6 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 3
  6 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 2
  6 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 3
  6 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 2
  6 months Post-Oxbryta: Missing | 187
  9 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 44
  9 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 21
  9 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 1
  9 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 2
  9 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 3
  9 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 1
  9 months Post-Oxbryta: Missing | 193
  12 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 50
  12 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 22
  12 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 2
  12 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 1
  12 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 2
  12 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 2
  12 months Post-Oxbryta: Missing | 186
  18 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 60
  18 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 29
  18 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 5
  18 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 0
  18 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 3
  18 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 3
  18 months Post-Oxbryta: Missing | 165
  24 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 55
  24 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 22
  24 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 3
  24 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 2
  24 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 1
  24 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 2
  24 months Post-Oxbryta: Missing | 180
  30 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 53
  30 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 21
  30 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 1
  30 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 4
  30 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 1
  30 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 1
  30 months Post-Oxbryta: Missing | 184
  36 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 39
  36 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 15
  36 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 4
  36 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 1
  36 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 1
  36 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 2
  36 months Post-Oxbryta: Missing | 203
  42 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 42
  42 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 12
  42 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 5
  42 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 0
  42 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 3
  42 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 1
  42 months Post-Oxbryta: Missing | 202
  48 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 33
  48 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 10
  48 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 4
  48 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 1
  48 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 5
  48 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 0
  48 months Post-Oxbryta: Missing | 212
  54 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 23
  54 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 6
  54 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 3
  54 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 0
  54 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 3
  54 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 2
  54 months Post-Oxbryta: Missing | 228
  60 months Post-Oxbryta: G1 - GFR >=90 mL/min per 1.73 m^2 | 7
  60 months Post-Oxbryta: G2 - GFR 60 to 89 mL/min per 1.73 m^2 | 1
  60 months Post-Oxbryta: G3a - GFR 45 to 59 mL/min per 1.73 m^2 | 1
  60 months Post-Oxbryta: G3b - GFR 30 to 44 mL/min per 1.73 m^2 | 0
  60 months Post-Oxbryta: G4 - GFR 15 to 29 mL/min per 1.73 m^2 | 0
  60 months Post-Oxbryta: G5 - GFR < 15 mL/min per 1.73 m^2 or treatment by dialysis | 0
  60 months Post-Oxbryta: Missing | 256

12. Primary Outcome: Number of Participants With SCD Complications
Description: SCD complications included acute pain crisis, acute chest syndrome (ACS), priapism, stroke, chronic or end stage kidney disease iron overload, leg ulcers, cardiac malfunction and pulmonary hypertension (PH) and RBC transfusions.
Time Frame: From date of first Oxbryta treatment through the end of study (up to Month 60)
Population: Safety analysis set (SAS) included all participants in the FAS who received at least one dose of Oxbryta including participants who had received at least one dose of Oxbryta in C5341018 (NCT04930328) (RETRO) study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 260
Participants | 205

13. Primary Outcome: Number of Participants With Treatment Initiation or Modification of SCD-related Medications
Description: Number of participants with treatment initiation or modification of SCD related medications is reported in this outcome measure.
Time Frame: From date of first Oxbryta treatment through the end of study (up to Month 60)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 260
Participants | 259

14. Primary Outcome: Number of Participants With Red Blood Cell (RBC) Transfusions
Description: Number of participants with RBC transfusions is reported in this outcome measure.
Time Frame: From date of first Oxbryta treatment through the end of study (up to Month 60)
Population: SAS included all participants in the FAS who received at least one dose of Oxbryta including participants who had received at least one dose of Oxbryta in C5341018 (NCT04930328) (RETRO) study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 260
Participants | 172

15. Primary Outcome: Number of Participants According to Responses to Patient Global Impression of Change (PGIC) at Month 3 Through Month 60
Description: PGIC was a single question that reflected a participant's or caregiver's belief about the effectiveness of treatment with Oxbryta on a 7-point scale depicting a participant's rating of overall improvement. Participants/caregivers rated their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse".
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 48
Participants
  Month 3: number analyzed (Participants) | 10
  Month 3: Very much improved | 1
  Month 3: Much improved | 2
  Month 3: Minimally improved | 3
  Month 3: No change | 4
  Month 3: Minimally worse | 0
  Month 3: Much worse | 0
  Month 3: Very much worse | 0
  Month 6: number analyzed (Participants) | 22
  Month 6: Very much improved | 4
  Month 6: Much improved | 6
  Month 6: Minimally improved | 6
  Month 6: No change | 5
  Month 6: Minimally worse | 0
  Month 6: Much worse | 1
  Month 6: Very much worse | 0
  Month 9: number analyzed (Participants) | 30
  Month 9: Very much improved | 6
  Month 9: Much improved | 6
  Month 9: Minimally improved | 8
  Month 9: No change | 10
  Month 9: Minimally worse | 0
  Month 9: Much worse | 0
  Month 9: Very much worse | 0
  Month 12: number analyzed (Participants) | 37
  Month 12: Very much improved | 2
  Month 12: Much improved | 12
  Month 12: Minimally improved | 8
  Month 12: No change | 15
  Month 12: Minimally worse | 0
  Month 12: Much worse | 0
  Month 12: Very much worse | 0
  Month 18: number analyzed (Participants) | 41
  Month 18: Very much improved | 4
  Month 18: Much improved | 17
  Month 18: Minimally improved | 11
  Month 18: No change | 7
  Month 18: Minimally worse | 2
  Month 18: Much worse | 0
  Month 18: Very much worse | 0
  Month 24: number analyzed (Participants) | 42
  Month 24: Very much improved | 3
  Month 24: Much improved | 14
  Month 24: Minimally improved | 9
  Month 24: No change | 13
  Month 24: Minimally worse | 1
  Month 24: Much worse | 1
  Month 24: Very much worse | 1
  Month 30: number analyzed (Participants) | 42
  Month 30: Very much improved | 6
  Month 30: Much improved | 12
  Month 30: Minimally improved | 11
  Month 30: No change | 11
  Month 30: Minimally worse | 1
  Month 30: Much worse | 1
  Month 30: Very much worse | 0
  Month 36: number analyzed (Participants) | 39
  Month 36: Very much improved | 4
  Month 36: Much improved | 12
  Month 36: Minimally improved | 16
  Month 36: No change | 5
  Month 36: Minimally worse | 2
  Month 36: Much worse | 0
  Month 36: Very much worse | 0
  Month 42: Very much improved | 8
  Month 42: Much improved | 11
  Month 42: Minimally improved | 17
  Month 42: No change | 11
  Month 42: Minimally worse | 1
  Month 42: Much worse | 0
  Month 42: Very much worse | 0
  Month 48: number analyzed (Participants) | 36
  Month 48: Very much improved | 1
  Month 48: Much improved | 17
  Month 48: Minimally improved | 9
  Month 48: No change | 7
  Month 48: Minimally worse | 1
  Month 48: Much worse | 0
  Month 48: Very much worse | 1
  Month 54: number analyzed (Participants) | 14
  Month 54: Very much improved | 0
  Month 54: Much improved | 5
  Month 54: Minimally improved | 3
  Month 54: No change | 6
  Month 54: Minimally worse | 0
  Month 54: Much worse | 0
  Month 54: Very much worse | 0
  Month 60: number analyzed (Participants) | 2
  Month 60: Very much improved | 0
  Month 60: Much improved | 2
  Month 60: Minimally improved | 0
  Month 60: No change | 0
  Month 60: Minimally worse | 0
  Month 60: Much worse | 0
  Month 60: Very much worse | 0

16. Primary Outcome: Number of Participants According to Responses to Clinical Global Impression of Change (CGIC) at Month 3 Through Month 60
Description: CGIC was a brief, stand-alone assessment of the clinician's view of the participant's global functioning prior to and after initiating Oxbryta. The CGI provided an overall clinician-determined summary measure that took into account all available information, including a knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. Participants rated their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," "very much worse," or "not assessed".
Time Frame: Month 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 30
Participants
  Month 3: number analyzed (Participants) | 4
  Month 3: Very much improved | 1
  Month 3: Much improved | 1
  Month 3: Minimally improved | 0
  Month 3: No change | 2
  Month 3: Minimally worse | 0
  Month 3: Much worse | 0
  Month 3: Very much worse | 0
  Month 3: Not assessed | 0
  Month 6: number analyzed (Participants) | 14
  Month 6: Very much improved | 1
  Month 6: Much improved | 1
  Month 6: Minimally improved | 6
  Month 6: No change | 5
  Month 6: Minimally worse | 1
  Month 6: Much worse | 0
  Month 6: Very much worse | 0
  Month 6: Not assessed | 0
  Month 9: number analyzed (Participants) | 19
  Month 9: Very much improved | 3
  Month 9: Much improved | 4
  Month 9: Minimally improved | 7
  Month 9: No change | 5
  Month 9: Minimally worse | 0
  Month 9: Much worse | 0
  Month 9: Very much worse | 0
  Month 9: Not assessed | 0
  Month 12: number analyzed (Participants) | 20
  Month 12: Very much improved | 1
  Month 12: Much improved | 4
  Month 12: Minimally improved | 7
  Month 12: No change | 7
  Month 12: Minimally worse | 0
  Month 12: Much worse | 0
  Month 12: Very much worse | 0
  Month 12: Not assessed | 1
  Month 18: number analyzed (Participants) | 29
  Month 18: Very much improved | 6
  Month 18: Much improved | 7
  Month 18: Minimally improved | 6
  Month 18: No change | 9
  Month 18: Minimally worse | 1
  Month 18: Much worse | 0
  Month 18: Very much worse | 0
  Month 18: Not assessed | 0
  Month 24: number analyzed (Participants) | 27
  Month 24: Very much improved | 3
  Month 24: Much improved | 13
  Month 24: Minimally improved | 6
  Month 24: No change | 2
  Month 24: Minimally worse | 2
  Month 24: Much worse | 0
  Month 24: Very much worse | 0
  Month 24: Not assessed | 1
  Month 30: number analyzed (Participants) | 19
  Month 30: Very much improved | 2
  Month 30: Much improved | 2
  Month 30: Minimally improved | 9
  Month 30: No change | 5
  Month 30: Minimally worse | 1
  Month 30: Much worse | 0
  Month 30: Very much worse | 0
  Month 30: Not assessed | 0
  Month 36: number analyzed (Participants) | 20
  Month 36: Very much improved | 1
  Month 36: Much improved | 8
  Month 36: Minimally improved | 6
  Month 36: No change | 4
  Month 36: Minimally worse | 0
  Month 36: Much worse | 0
  Month 36: Very much worse | 1
  Month 36: Not assessed | 0
  Month 42: Very much improved | 0
  Month 42: Much improved | 12
  Month 42: Minimally improved | 10
  Month 42: No change | 8
  Month 42: Minimally worse | 0
  Month 42: Much worse | 0
  Month 42: Very much worse | 0
  Month 42: Not assessed | 0
  Month 48: number analyzed (Participants) | 21
  Month 48: Very much improved | 2
  Month 48: Much improved | 1
  Month 48: Minimally improved | 10
  Month 48: No change | 6
  Month 48: Minimally worse | 1
  Month 48: Much worse | 0
  Month 48: Very much worse | 0
  Month 48: Not assessed | 1
  Month 54: number analyzed (Participants) | 6
  Month 54: Very much improved | 0
  Month 54: Much improved | 0
  Month 54: Minimally improved | 2
  Month 54: No change | 4
  Month 54: Minimally worse | 0
  Month 54: Much worse | 0
  Month 54: Very much worse | 0
  Month 54: Not assessed | 0
  Month 60: number analyzed (Participants) | 2
  Month 60: Very much improved | 1
  Month 60: Much improved | 1
  Month 60: Minimally improved | 0
  Month 60: No change | 0
  Month 60: Minimally worse | 0
  Month 60: Much worse | 0
  Month 60: Very much worse | 0
  Month 60: Not assessed | 0

17. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) According to Severity
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and other important medical events. Severity was classified using common terminology criteria for adverse events (CTCAE), version 5.0, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe. Mild - SAEs does not interfere with participant's usual function b) moderate - SAEs interferes to some extent with participant's usual function c) severe - SAEs interferes significantly with participant's usual function.
Time Frame: From date of first Oxbryta treatment up to end of study (up to Month 60)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants with SCD and treated with voxelotor as prescribed by their physician were included, with no pre-defined treatment regimen required.
Arm/Group | All Participants
Number analyzed (Participants) | 260
Participants
  Mild | 8
  Moderate | 55
  Severe | 87

18. Primary Outcome: Number of Participants With Adverse Events (AEs) According to Severity
Description: An AE was any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. Severity was classified using CTCAE, version 5.0, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe. AEs are classified according to the severity in 3 categories a) mild - AEs does not interfere with participant's usual function b) moderate - AEs interferes to some extent with participant's usual function c) severe - AEs interferes significantly with participant's usual function. AEs included both SAEs and non-SAEs.
Time Frame: From date of first Oxbryta treatment up to end of study (up to Month 60)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 260
Participants
  Mild | 28
  Moderate | 83
  Severe | 99

19. Primary Outcome: Number of Participants With AEs Leading to Dose Modification or Discontinuation of Oxbryta
Description: An AE was any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Number of participants with AEs leading to dose modification or discontinuation of Oxbryta were reported in this outcome measure.
Time Frame: From date of first Oxbryta treatment up to end of study (up to Month 60)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 260
Participants | 7

20. Primary Outcome: Number of Participants With Positive Pregnancy Test and Fertility Complications
Description: Number of participants with positive pregnancy test and fertility complications were reported in this outcome measure.
Time Frame: From date of first Oxbryta treatment up to end of study (up to Month 60)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 260
Participants | 7

21. Other Pre Specified Outcome: Change in Number of Outpatient Visits From Pre-Oxbryta Treatment
Description: Outpatient visits (including infusion center, acute care, or telemedicine visit) were planned to be analyzed.
Time Frame: From date of first Oxbryta treatment through the end of study (up to Month 60)
Population: Data for this outcome measure was not collected due to premature termination of the study. Only limited efficacy data to support the benefit-risk evaluation of Oxbryta was collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

22. Other Pre Specified Outcome: Change in Number of Emergency Department (ED) Visits From Pre-Oxbryta Treatment
Description: ED visits were planned to be analyzed in this outcome measure.
Time Frame: From date of first Oxbryta treatment through the end of study (up to Month 60)
Population: as for outcome 21
Arm/Group | All Participants
Number analyzed (Participants) | 0

23. Other Pre Specified Outcome: Change in Number of Hospitalizations From Pre-Oxbryta Treatment
Description: Number of hospitalizations were planned to be analyzed.
Time Frame: From date of first Oxbryta treatment through the end of study (up to Month 60)
Population: as for outcome 21
Arm/Group | All Participants
Number analyzed (Participants) | 0

24. Other Pre Specified Outcome: Change in Home Oxygen Supplementation From Pre-Oxbryta Treatment
Time Frame: From date of first Oxbryta treatment through the end of study (up to Month 60)
Population: as for outcome 21
Arm/Group | All Participants
Number analyzed (Participants) | 0

25. Other Pre Specified Outcome: Number of Participants With Renal Dialysis
Time Frame: From date of first Oxbryta treatment through the end of study (up to Month 60)
Population: as for outcome 21
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From date of first Oxbryta treatment up to end of study (up to Month 60)
Description: Same event may occur as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. SAS included all participants in the FAS who received at least one dose of Oxbryta including participants who had received at least one dose of Oxbryta in C5341018 (NCT04930328) (RETRO) study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 6/260
Serious Adverse Events (participants affected / at risk) | 150/260
Other Adverse Events (participants affected / at risk) | 185/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=260)
Anaemia (Blood and lymphatic system disorders) | 4
Aplastic anaemia (Blood and lymphatic system disorders) | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Hypersplenism (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 131
Splenomegaly (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Pulmonary valve incompetence (Cardiac disorders) | 1
Sickle cell anaemia (Congenital, familial and genetic disorders) | 8
Goitre (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Tooth impacted (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden death (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Abdominal wall abscess (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 6
Clostridium difficile colitis (Infections and infestations) | 1
Corynebacterium bacteraemia (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Mycobacterial infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 19
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Delayed haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Epstein-Barr virus test positive (Investigations) | 1
Staphylococcus test positive (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Iron overload (Metabolism and nutrition disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 8
Cerebrovascular accident (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Middle cerebral artery stroke (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Psychogenic seizure (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Hallucination (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 3
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 59
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Brachiocephalic artery occlusion (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 5
Jugular vein occlusion (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Subclavian vein occlusion (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=260)
Anaemia (Blood and lymphatic system disorders) | 1
Haemolysis (Blood and lymphatic system disorders) | 1
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 154
Atrial thrombosis (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Sickle cell anaemia (Congenital, familial and genetic disorders) | 9
Ophthalmic artery aneurysm (Eye disorders) | 1
Retinopathy (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 30
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 47
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 38
Pancreatitis acute (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Drug ineffective (General disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 5
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 8
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Blood bilirubin unconjugated increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Iron overload (Metabolism and nutrition disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 13
Cerebral infarction (Nervous system disorders) | 1
Headache (Nervous system disorders) | 40
Intracranial aneurysm (Nervous system disorders) | 1
End stage renal disease (Renal and urinary disorders) | 2
Priapism (Reproductive system and breast disorders) | 1
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 16
Skin ulcer (Skin and subcutaneous tissue disorders) | 4
Deep vein thrombosis (Vascular disorders) | 5
Superficial vein thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
For outcome measure 9, the terminology used for other: small, medium, and large were entered by sites to describe the severity or amount but is not clinically precise and should be interpreted cautiously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT04930445/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT04930445/SAP_001.pdf